CLINICAL TRIAL: NCT06913322
Title: Flush Versus Standard Distance From Saphenofemoral Junction in Endovenous Laser Ablation of Great Saphenous Vein
Acronym: fEVLA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Abdullah Yahya Mohamed Fouda, doctor, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KFSIRB200-278; MUka12 (Other: Cairo university)
Record Dates: First submitted 2025-03-23; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Varicose Veins Leg
Keywords: laser ablation; flush; standard distance
MeSH Terms: conditions — Blushing

STUDY DESIGN:
Intervention Model Description: endovenous laser ablation of lower limb varicose veins
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- flush EVLA (Active Comparator): The fiber tip was positioned in fEVLA group Flush at SFJ
  Interventions: Procedure: flush endovenous laser ablation of great saphenous vein
- standard EVLA (Active Comparator): The fiber tip was positioned in sEVLA group 2 cm distal to SFJ
  Interventions: Procedure: standard endovenous laser ablation of great saphenous vein

INTERVENTIONS:
Procedure: flush endovenous laser ablation of great saphenous vein — A 4 French sheath is advanced over the wire and positioned in the great saphenous vein below knee. Diode laser (SmartM; Lasotronix) with a 600-mm radial fiber catheter was used. The tip of the laser was be placed flush at saphenofemoral junction.
  Arms: flush EVLA
Procedure: standard endovenous laser ablation of great saphenous vein — A 4 French sheath is advanced over the wire and positioned in the great saphenous vein below knee. Diode laser (SmartM; Lasotronix) with a 600-mm radial fiber catheter was used. The tip of the laser was be placed 2 cm distal to saphenofemoral junction.
  Arms: standard EVLA

SUMMARY:
Varicose veins of the great saphenous vein (GSV) are a prevalent venous disorder, with higher incidence in women. They cause swelling, pain, ulcers, eczema, and phlebitis, impacting patients' occupational performance and quality of life. Endovenous laser ablation (EVLA) has been supplanted by high-level laser surgery (HLS) as the primary treatment for incompetent GSVs. EVLA uses laser energy to generate heat, altering or inactivating proteins and enzymes within the vessel wall. Occlusion rates are shown to be around 95% after one year. However, the influence of the untreated proximal segment adjacent to the sapheno-femoral junction (SFJ) on reflux and recurrence is ambiguous. Contemporary laser fibers, such as radially emitting fibers, can reduce postoperative discomfort and improve outcomes. However, data on the safety and long-term outcomes of flush ablation compared to standard ablation remains insufficient.

DETAILED DESCRIPTION:
Varicose veins of the great saphenous vein (GSV) represent one of the most prevalent venous disorders, with a higher incidence in women compared to men. The manifestations of varicose veins include not only swelling and pain in the lower extremities but are frequently associated with ulcers, eczema, phlebitis, and other detrimental effects, resulting in an irreversible impact on patients' occupational performance and quality of life. To enhance this, it is essential to investigate appropriate treatments for clinical implementation (3). Current guidelines indicate that EVLA and other endovenous thermal ablation techniques have supplanted HLS as the primary treatment for incompetent saphenous veins, due to their demonstrated efficacy in numerous countries. In the EVLA treatment, laser energy is introduced into the lumen of the blood vessel, generating heat that alters or inactivates the proteins and enzymes within the vessel wall. Following the destruction of the vein wall's structure, the vein exhibits fibrosis, resulting in the contraction and permanent occlusion of the blood vessels. Endovenous laser ablation (EVLA) is an efficacious technique for addressing incompetent great saphenous veins (GSV) (5, 6, 7). Occlusion rates were shown to attain approximately 95% after one year (5). Notwithstanding favorable outcomes regarding the occlusion rate, the influence of the untreated proximal segment adjacent to the sapheno-femoral junction (SFJ) on the onset of reflux and recurrence following thermal ablation remains ambiguous (8, 9, 10, 11). Increased incidences of stump reflux following EVLA have been documented in comparison to high ligation and stripping (8, 9). Flessenkämper et al. demonstrated a significantly higher incidence of reflux from the SFJ into the GSV following EVLA alone compared to high ligation and stripping (HL/S) and HL plus EVLA (8). Rass et al. reported a 17.8% incidence of reflux in the GSV stump following EVLA and a 1.3% incidence after HL/S (9). The authors consequently reported a greater incidence of recurrent varicose veins in the groin compared to high ligation/stripping after five years (9). Contemporary laser fibers, such as radially emitting fibers, can diminish postoperative discomfort and enhance outcomes (12, 13). A modified radial fiber emits laser energy in two distinct rings radially around the tip. This is believed to produce a more uniform thermal effect on the venous wall, resulting in reduced pain and bruising post-procedure (14). These fibers facilitate the ablation of the GSV near the SFJ and may yield results comparable to high ligation (15). A comparable effect can be achieved with the 1-ring fiber, exhibiting a slightly elevated linear energy density (LEED) at the junction with the deep vein. This study will utilize the 2-ring fiber, as we favor a marginally diminished LEED at the tip to mitigate the risk of injury to the deep vein. Regrettably, data regarding the safety and long-term outcomes of flush ablation in comparison to standard ablation remain insufficient.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years.
* patients with CEAP classes C2 to C6
* primary great saphenous vein insufficiency with at least 0.5 seconds of reflux in the standing position on color Doppler ultrasound.

Exclusion Criteria:

* deep or superficial venous thrombosis
* previous treatment of the varicose veins
* severe infection in the ipsilateral lower limb
* GSV diameter more than15 mm or less than 3 mm
* ipsilateral lower limb arterial stenosis or occlusion;
* pregnancy or breastfeeding;
* iliac vein compression syndrome.
* congenital venous anomalies
* allergy to lidocaine
* Debilitating systemic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-01-21 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
occlusion rate | 1 year
  1-percentage of treated veins that remain closed or occluded (blocked) following the EVLA. It is an important measure of the treatment's effectiveness in permanently sealing the vein, preventing blood flow through ablated area.
endovenous heat induced thrombosis | 1 year
  formation of a blood clot at saphenofemoral junction caused by heat from endovenous laser ablation of great saphenous vein

SECONDARY OUTCOMES:
complications | 1 year
  Procedure-related complications, such as deep venous thrombosis in locations other than the SFJ or CFV, superficial vein thrombosis, pulmonary embolism, allergy, sensory disturbance in the groin region, bleeding, and infection

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafrelsheikh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gauw SA, Lawson JA, van Vlijmen-van Keulen CJ, Pronk P, Gaastra MT, Mooij MC. Five-year follow-up of a randomized, controlled trial comparing saphenofemoral ligation and stripping of the great saphenous vein with endovenous laser ablation (980 nm) using local tumescent anesthesia. J Vasc Surg. 2016 Feb;63(2):420-8. doi: 10.1016/j.jvs.2015.08.084. Epub 2015 Oct 23. PMID 26602795
- [Background] Hirokawa M, Ogawa T, Sugawara H, Shokoku S, Sato S. Comparison of 1470 nm Laser and Radial 2ring Fiber with 980 nm Laser and Bare-Tip Fiber in Endovenous Laser Ablation of Saphenous Varicose Veins: A Multicenter, Prospective, Randomized, Non-Blind Study. Ann Vasc Dis. 2015;8(4):282-9. doi: 10.3400/avd.oa.15-00084. Epub 2015 Sep 9. PMID 26730252
- [Background] Pannier F, Rabe E, Rits J, Kadiss A, Maurins U. Endovenous laser ablation of great saphenous veins using a 1470 nm diode laser and the radial fibre--follow-up after six months. Phlebology. 2011 Feb;26(1):35-9. doi: 10.1258/phleb.2010.009096. Epub 2010 Dec 9. PMID 21148467
- [Background] Doganci S, Demirkilic U. Comparison of 980 nm laser and bare-tip fibre with 1470 nm laser and radial fibre in the treatment of great saphenous vein varicosities: a prospective randomised clinical trial. Eur J Vasc Endovasc Surg. 2010 Aug;40(2):254-9. doi: 10.1016/j.ejvs.2010.04.006. Epub 2010 May 23. PMID 20547079
- [Background] Theivacumar NS, Darwood R, Gough MJ. Neovascularisation and recurrence 2 years after varicose vein treatment for sapheno-femoral and great saphenous vein reflux: a comparison of surgery and endovenous laser ablation. Eur J Vasc Endovasc Surg. 2009 Aug;38(2):203-7. doi: 10.1016/j.ejvs.2009.03.031. Epub 2009 Jun 12. PMID 19524460
- [Background] O'Donnell TF, Balk EM, Dermody M, Tangney E, Iafrati MD. Recurrence of varicose veins after endovenous ablation of the great saphenous vein in randomized trials. J Vasc Surg Venous Lymphat Disord. 2016 Jan;4(1):97-105. doi: 10.1016/j.jvsv.2014.11.004. Epub 2015 Apr 11. PMID 26946904
- [Background] Rass K, Frings N, Glowacki P, Graber S, Tilgen W, Vogt T. Same Site Recurrence is More Frequent After Endovenous Laser Ablation Compared with High Ligation and Stripping of the Great Saphenous Vein: 5 year Results of a Randomized Clinical Trial (RELACS Study). Eur J Vasc Endovasc Surg. 2015 Nov;50(5):648-56. doi: 10.1016/j.ejvs.2015.07.020. Epub 2015 Aug 28. PMID 26319476
- [Background] Flessenkamper I, Hartmann M, Hartmann K, Stenger D, Roll S. Endovenous laser ablation with and without high ligation compared to high ligation and stripping for treatment of great saphenous varicose veins: Results of a multicentre randomised controlled trial with up to 6 years follow-up. Phlebology. 2016 Feb;31(1):23-33. doi: 10.1177/0268355514555547. Epub 2014 Oct 22. PMID 25342648
- [Background] Disselhoff BC, der Kinderen DJ, Kelder JC, Moll FL. Five-year results of a randomised clinical trial of endovenous laser ablation of the great saphenous vein with and without ligation of the saphenofemoral junction. Eur J Vasc Endovasc Surg. 2011 May;41(5):685-90. doi: 10.1016/j.ejvs.2010.12.014. Epub 2011 Feb 18. PMID 21333560
- [Background] Pannier F, Rabe E, Maurins U. First results with a new 1470-nm diode laser for endovenous ablation of incompetent saphenous veins. Phlebology. 2009 Feb;24(1):26-30. doi: 10.1258/phleb.2008.008038. PMID 19155338
- [Background] Lawaetz M, Serup J, Lawaetz B, Bjoern L, Blemings A, Eklof B, Rasmussen L. Comparison of endovenous ablation techniques, foam sclerotherapy and surgical stripping for great saphenous varicose veins. Extended 5-year follow-up of a RCT. Int Angiol. 2017 Jun;36(3):281-288. doi: 10.23736/S0392-9590.17.03827-5. Epub 2017 Feb 17. PMID 28217989
- [Background] Castro-Ferreira R, Quelhas MJ, Freitas A, Vidoedo J, Silva EA, Marinho A, Abreu R, Coelho A, Dias PG, Sampaio SM. Vascular training does matter in the outcomes of saphenous high ligation and stripping. J Vasc Surg Venous Lymphat Disord. 2019 Sep;7(5):732-738. doi: 10.1016/j.jvsv.2019.01.060. Epub 2019 May 5. PMID 31068278
- [Background] Carroll C, Hummel S, Leaviss J, Ren S, Stevens JW, Everson-Hock E, Cantrell A, Stevenson M, Michaels J. Clinical effectiveness and cost-effectiveness of minimally invasive techniques to manage varicose veins: a systematic review and economic evaluation. Health Technol Assess. 2013 Oct;17(48):i-xvi, 1-141. doi: 10.3310/hta17480. PMID 24176098
- [Background] Carradice D, Mekako AI, Mazari FA, Samuel N, Hatfield J, Chetter IC. Randomized clinical trial of endovenous laser ablation compared with conventional surgery for great saphenous varicose veins. Br J Surg. 2011 Apr;98(4):501-10. doi: 10.1002/bjs.7394. Epub 2011 Jan 31. PMID 21283981
- [Background] Tauraginskii RA, Lurie F, Agalarov R, Simakov S, Borsuk D. Blood flow from competent tributaries is likely contributor to distally increasing reflux volume in incompetent great saphenous vein. J Vasc Surg Venous Lymphat Disord. 2022 Jan;10(1):69-74. doi: 10.1016/j.jvsv.2021.04.010. Epub 2021 May 4. PMID 33957280